CLINICAL TRIAL: NCT06401694
Title: Evaluating the Impact and Sustainability of Enhanced Home-delivered Meal Program Services on Older Adults' Health and Well-being
Brief Title: Evaluating an Enhanced Home-delivered Meal Program on Older Adults' Health and Well-being
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Meals on Wheels Rhode Island (MOWRI) (Unknown)
Responsible Party: Principal Investigator, Caitlin Caspi, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-073-910
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diet, Healthy; Food Insecurity; Loneliness; Quality of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced (Experimental): Home-delivered meals plus Community Health Worker Calls and supplemental grocery bags
  Interventions: Other: Home-delivered meals; Other: Wellness check and socialization visit; Behavioral: Community Health Worker calls; Other: Supplemental grocery bag
- Usual care (Active Comparator): Home-delivered meals
  Interventions: Other: Home-delivered meals; Other: Wellness check and socialization visit

INTERVENTIONS:
Other: Home-delivered meals — Delivery of prepared meals compliant with Older Americans Act nutrition programs guidelines
Other: Wellness check and socialization visit — At-home delivery with opportunity for driver observation and interaction
Behavioral: Community Health Worker calls — Calls from a certified Community Health Worker (CHW) to assess needs, identify gaps in care and resources, and then support health and resource coordination
  Arms: Enhanced
Other: Supplemental grocery bag — Monthly delivery of a grocery bag containing a variety of nutritionally balanced foods and educational materials
  Arms: Enhanced

SUMMARY:
Meals on Wheels of Rhode Island (MOWRI), in partnership with the University of Connecticut (UConn), will implement and evaluate an enhanced version of its Home-Delivered Meals Program (HDMP). The project goal is to implement and test the effectiveness of an enhanced Home-Delivered Meals (HDM) service delivery approach. The enhanced approach includes community health worker (CHW) interactions and supplemental healthy grocery bags to address diet quality, food and nutrition security, loneliness, and health-related quality of life for older adults. MOWRI participants at the highest nutritional risk will be randomized to receive standard or enhanced services in order to test the effect of the intervention on health-related outcomes. Anticipated outcomes for individuals receiving enhanced services are improvements in measures of diet quality, food and nutrition security, loneliness, and health-related quality of life compared with those receiving standard HDM services.

DETAILED DESCRIPTION:
The purpose of the research study is to understand the effectiveness of an enhanced Home-Delivered Meals Program (HDMP) on the health-quality of life for older adults. Specifically, the investigators will study the effectiveness of an enhanced HDMP service delivery approach that includes community health worker interactions and supplemental healthy grocery bags to address diet quality, food and nutrition security, loneliness, and health-related quality of life, compared to HDMP only. The research will take place among individuals receiving meals from Meals on Wheels Rhode Island (MOWRI). This is a pragmatic randomized controlled trial with the following objectives: 1) to develop a protocol for CHW engagement (assessment, intervention, and follow-up) with participants; 2) to implement the enhanced home delivered meals (HDM) intervention to MOWRI clients at the highest nutritional risk; 3) to evaluate the impact of the enhanced program on diet quality, food and nutrition security, loneliness, and HRQOL in a randomized study; 4) to evaluate program sustainability measures and implement process improvements to increase sustainability; 5) to disseminate program resources that will allow the program to replicate to other HDM programs; and 6) to share evaluation results with key community, policy, and academic partners. Up to 1640 participants who are individuals receiving meals from Meals on Wheels Rhode Island (MOWRI) and are at a high nutritional risk. The outcome measures are diet quality (primary outcome), food security, nutrition security, subjective isolation / loneliness, health-related quality of life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

* Adults who are eligible for Title III - funded Meals on Wheels assistance
* Can read and speak Spanish or English
* Are nutritionally at risk as determined by the Nutrition Risk Assessment
* Reside in the state of Rhode Island

Exclusion Criteria:

* Cognitive or physical limitations that prevent an individual from giving consent, as assessed by normal interactions by intake staff or study team
* Cognitive or physical limitations that prevent an individual from participating in intervention or evaluation activities, as assessed by normal interactions intake staff or study team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1640 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Diet Quality | 12 weeks
  Dietary Screening Tool (DST); Minimum value (0) indicates lowest possible score; Maximum value (100) indicates highest possible score

SECONDARY OUTCOMES:
Food Security | 12 weeks
  U.S. Household Food Security Survey Module: Six-Item Short Form; Minimum value (0) indicates high food security; Maximum value (6) indicates very low food security
Nutrition Security | 12 weeks
  2-item Nutrition Security Screener (NSS); participants responding (a) very hard, (b) hard, or (c) somewhat hard to the first question will be designated as nutrition insecure.
Loneliness | 12 weeks
  University of California, Los Angeles 3-Item Loneliness Scale; Minimum value (3) indicates low feelings of loneliness; Maximum value (9) indicates high feelings of loneliness
Health-Related Quality of Life | 12 weeks
  The Centers for Disease Control and Prevention's Health-Related Quality of Life 4-question core modules, called the "Healthy Days Measures"; The unhealthy days index is calculated by summing the number of physically and mentally unhealthy days, capped at 30 total days.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Caspi, ScD, Principal Investigator — University of Connecticut; Kim Gans, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa da Silva IL, Gans KM, Thomas KS, Gutman R, Tyler B, Ray S, Grady M, DeFelice S, Hussein M, Lusi A, Caspi CE. A study protocol for a randomized controlled trial evaluating the impact of adding community health worker coaching calls and healthy grocery bag deliveries to a Meals on Wheels home-delivered meal program for homebound older adults in Rhode Island. BMC Public Health. 2025 Oct 1;25(1):3285. doi: 10.1186/s12889-025-24080-6. PMID 41034808